CLINICAL TRIAL: NCT06277739
Title: Brain Effect Mechanism of Spinal Manipulative Therapy on Lumbar Disc Herniation Analgesia Based on Multimodal Magnetic Resonance Imaging
Brief Title: Brain Effect Mechanism of Spinal Manipulative Therapy on LDH Analgesia Based on Multimodal MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhou Xingchen (Other)
Responsible Party: Sponsor-Investigator, Zhou Xingchen, Prof., The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20220117020315695
Record Dates: First submitted 2024-02-14; First posted 2024-02-26 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Lumbar Disc Herniation
Keywords: Lumbar Disc Herniation; Spinal Manipulative Therapy; MRI
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group1 (Spinal Manipulation Therapy) (Experimental): The participant was placed in a side-lying position facing the clinician with the more painful side facing upward. The clinician passively flexed the participant's hips and knees to induce lumbar spine flexion until they felt the spinous process of the affected lumbar vertebrae begin to move. Next, the clinician passively rotated the participant's torso opposite to the side they were lying on until they felt rotation in the vertebra above the suspected lesion. The clinician applied a rapid thrust to the shoulder (anterior to posterior force) and pelvis (posterior to anterior force) resulting in a rotation force couple on the hypomobile segment.
  Interventions: Procedure: Spinal Manipulative Therapy
- Group2 Sham Laser Treatment) (Placebo Comparator): The laser manufacturer (MedX Health Corp) provided a MedX 1100 system that did not deliver any significant amount of light energy or heat but otherwise appeared operational to participants and clinicians. The sham laser was delivered over the painful region with the study participant positioned as described for spinal manipulation and spinal mobilization treatments.
  Interventions: Other: Sham Laser Treatment
- Group3 (healthy controls) (No Intervention)

INTERVENTIONS:
Procedure: Spinal Manipulative Therapy — The participant was placed in a side-lying position facing the clinician with the more painful side facing upward. The clinician passively flexed the participant's hips and knees to induce lumbar spine flexion until they felt the spinous process of the affected lumbar vertebrae begin to move. Next, the clinician passively rotated the participant's torso opposite to the side they were lying on until they felt rotation in the vertebra above the suspected lesion. The clinician applied a rapid thrust to the shoulder (anterior to posterior force) and pelvis (posterior to anterior force) resulting in a rotation force couple on the hypomobile segment. If a cavitation (ie, an audible pop) occurred, the treatment was considered complete. If no cavitation was produced, the participant was repositioned and the manipulation was attempted again. A maximum of 2 attempts per side was permitted. If no cavitation was produced after the 4 attempts (ie, 2 per side), the treatment was considered complete.
  Arms: Group1 (Spinal Manipulation Therapy)
Other: Sham Laser Treatment — The laser manufacturer (MedX Health Corp) provided a MedX 1100 system that did not deliver any significant amount of light energy or heat but otherwise appeared operational to participants and clinicians. The sham laser was delivered over the painful region with the study participant positioned as described for spinal manipulation and spinal mobilization treatments.
  Arms: Group2 Sham Laser Treatment)

SUMMARY:
The clinical symptoms of Lumbar Disc Herniation (LDH) can be effectively ameliorated through Spinal Manipulative Therapy (SMT), which is closely linked to the brain's pain-regulating mechanisms. Magnetic Resonance Imaging (MRI) offers an objective and visual means to study how the brain orchestrates the characteristics of analgesic effects. From the perspective of multimodal MRI, the investigators applied functional MRI (fMRI) and Magnetic Resonance Spectrum (MRS) techniques to comprehensively evaluate the characteristics of the effects of SMT on the brain region of LDH from the aspects of brain structure, brain function and brain metabolism. This multimodal MRI technique provides a biological basis for the clinical application of SMT in LDH.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the diagnostic criteria for lumbar disc herniation, including protrusion types such as central, paracentral, far lateral, foraminal, and subarticular, with imaging findings that align with neurological localization.
* The age range for participants is 18 to 65 years, encompassing any gender, and they must be right-handed.
* Participants should be in the non-acute phase of the condition, experiencing mild to moderate pain and functional impairment, with the duration of symptoms exceeding 2 weeks.
* Participants should have a Visual Analog Scale (VAS) score greater than 4 and Japanese Orthopaedic Association (JOA) scores less than 15.
* Eligible participants must not have taken analgesics, neurotropic nutrition drugs, or sedatives in the past month and should not have undergone systemic treatment.
* Participants should not have received spinal manipulation or other physical therapies in the past month.
* Participants must voluntarily agree to participate in this study and have signed an informed consent form.

Exclusion Criteria:

* Patients with concurrent internal medicine or gynecological conditions known to cause lower back pain, such as nephritis, urinary stones, gynecological inflammations, and uterine abnormalities.
* Individuals with severe primary diseases impacting the cardiovascular, cerebrovascular, liver, or kidney systems.
* Those with neurogenic functional disorders, psychiatric conditions, a history of significant head trauma, or a history of unconsciousness.
* Individuals diagnosed with primary sciatica or dry sciatica.
* Those with lumbar spondylolisthesis.
* Patients suffering from lumbar tumors or tuberculosis.
* Individuals with severe osteoporosis or localized skin lesions in the lumbar area.
* Patients experiencing painful conditions beyond the lumbar region.
* Those with diseases characterized by structural changes in the brain.
* Individuals with impaired consciousness, severe visual or hearing impairments, speech disorders, or others who are unable to complete health assessments.
* Individuals with dental implants, metal stents, or other elements that may compromise MRI imaging.
* Those with a fear of MRI or other reasons that prevent undergoing MRI scans.
* Patients diagnosed with lumbar disc herniation but who are asymptomatic.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
visual analogue scale (VAS) | up to one month
  Pain intensity was evaluated by means of a visual analogue scale (VAS) [10-point visual analogue scale: 0 = no pain; 10 = very severe pain].
Japanese Orthopaedic Association Scores (JOA) | up to one months
  Japanese Orthopaedic Association Scores (JOA), ranging from 0 (worst) to 100 (best), was used to evaluate the clinical state.
Amplitude of Low-Frequency Fluctuation (ALFF) | up to one months
  The ALFF measures the activity of neurons in the brain that are not affected by external factors.
Regional Homogeneity (ReHo) | up to one months
  The ReHo measures the consistency of the local functional activities of the brain's various regions.
Functional Connectivity (FC) | up to one months
  The FC represents the strength Of functional connections between brain regions, and can reflect the temporal correlation between the Region Of Interest (ROI) and the whole brain networking function.
Magnetic Resonance Spectrum （MRS） | up to one month
  The MRS Is the only technology capable of non-invasive quantitative detection of brain substance changes.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-zhen Lv, Ph.D., Study Director — The Third School of Clinical Medicine, Zhejiang Chinese Medical University
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Zhou XC, Wu S, Wang KZ, Chen LH, Wei ZC, Li T, Hua ZH, Xia Q, Lyu ZZ, Lyu LJ. Impact of Spinal Manipulative Therapy on Brain Function and Pain Alleviation in Lumbar Disc Herniation: A Resting-State fMRI Study. Chin J Integr Med. 2025 Feb;31(2):108-117. doi: 10.1007/s11655-024-4205-7. Epub 2024 Dec 21. PMID 39707137